CLINICAL TRIAL: NCT03523429
Title: A Phase II, Open-label Study to Evaluate the Effect of Blinatumomab Administered During Consolidation to Reduce the Level of Minimal Residual Disease (MRD) Assessed Through Flow Cytometry in Adult Patients up to 55 Years of Age With High-risk Philadelphia Chromosome-negative (Ph-) Acute Lymphoblastic Leukaemia (ALL) With Good Response (MRD < 0.1%) After Induction Therapy
Brief Title: PETHEMA-BLIN-01/PET069014 (BLIN-01)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low rate of recruitment
Sponsor: PETHEMA Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PETHEMA-BLIN-01
Record Dates: First submitted 2018-05-01; First posted 2018-05-14 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Philadelphia Chromosome-negative or BCR-ABL-negative, CD19-positive ALL
MeSH Terms: interventions — blinatumomab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- blinatumomab (Experimental): blinatumomab administered during the early consolidation phase in patients ≤ 55 years with high-risk Philadelphia chromosome-negative (Ph-) acute lymphoblastic leukaemia (ALL) with MRD < 0.1% (< 1×10-3) after induction therapy.
  Interventions: Drug: blinatumomab

INTERVENTIONS:
Drug: blinatumomab — Blinatumomab is a bispecific monoclonal antibody designed to bind specifically to CD19, expressed on the surface of B-cells, and to CD3, expressed on the surface of T-cells. It activates endogenous T-cells by connecting the CD3 on the T-cell receptor complex (TCR) with the CD19 on the B-cells. The anti-tumour activity of blinatumomab does not depend on whether the T-cells carry a specific TCR or peptide antigens present in cancer cells, but it is polyclonal and independent of HLA on the target cells

SUMMARY:
The PETHEMA Spanish group treats patients with high-risk Philadelphia chromosome-negative ALL, aged 18 to 55 years, based on the MRD clearance as assessed by flow cytometry at a centralised evaluation centre. Patients with MRD < 0.1% (< 1×10-3) after induction and < 0.01% (< 1×10-4) after early consolidation are assigned to receive chemotherapy (late consolidation and maintenance).

Early consolidation chemotherapy consists of three cycles including high doses of MTX, ARA-C and ASP, together with vincristine and dexamethasone. The same therapy is repeated in the late consolidation period if MRD after early consolidation is < 0.01% (< 1×10-4). Maintenance therapy is then administered for up to 2 years from the CR date. These patients do not receive allo-HSCT if they maintain adequate MRD clearance.

Despite having adequate MRD clearance, a proportion of patients (around 25%) experience relapse, which makes other approaches necessary to try to decrease the relapse rate. Intensifying currently existing chemotherapy regimens is not likely to increase the cure rate and would likely significantly increase toxicity. The use of targeted immunotherapeutic agents such as blinatumomab, which has demonstrated efficacy and safety in patients with R/R ALL and in patients with ALL and MRD+, seems to be a promising option [30-33].

Therefore, it would be interesting to assess the potential efficacy of using blinatumomab in CR patients to reduce the MRD more frequently and more intensely during the early and late consolidation period. Our hypothesis is that blinatumomab will further reduce the level of MRD and this could lead to a decrease in the relapse rate in these patients.

This trial will replace the third early consolidation cycle with a cycle of blinatumomab, and the same will be done in the late consolidation period. We hope that this strategy will increase the extent of the MRD response and prevent relapses.

Moreover, and as a secondary objective, we will investigate the safety of blinatumomab administration after the administration of high-dose chemotherapy including MTX, ARA-C and ASP

DETAILED DESCRIPTION:
In the pre-phase, patients receive treatment according to routine clinical practice at Spanish sites, in accordance with the PETHEMA protocol for patients with high-risk ALL (ALL-AR-11), with: Prednisone (PDN) 60 mg/m2, PO or IV until complete characterisation of the ALL, for a maximum of 7 days, Triple intrathecal therapy, Methotrexate (MTX) 12 mg, ARA-C: 30 mg, Hydrocortisone 20 mg.

Standard induction chemotherapy that these patients receive according to routine clinical practice at Spanish sites, in accordance with the PETHEMA protocol for patients with high-risk ALL (ALL-AR-11), consists of: Vincristine (VCR) 1.5 mg/m2 (maximum dose 2 mg) IV days 1, 8, 15 and 22,Daunorubicin (DNR) 45 mg/m2 IV days 1, 8, 15 and 22, prednisone 60 mg/m2 per day, IV or PO, days 1 to 14,30 mg/m2 per day, IV or PO, days 15 to 21, 15 mg/m2 per day, IV or PO, days 21 to 28,E. coli L-asparaginase (L-ASP) (Kidrolase®) 10,000 IU/m2, IV, days 16-20, 23-27,Intrathecal TIT chemotherapy day 1* (if not administered in the pre-phase) and 22, Methotrexate (MTX) 12 mg, ARA-C: 30 mg, Hydrocortisone 20 mg, G-CSF (SC or IV) from day 15 until neutrophils > 1000/µl.

Following the administration of induction therapy, a bone marrow analysis will be performed with morphological, genetic and molecular study if necessary, with a centralised MRD determination by MFC. In the case of a complete morphological response and MRD < 0.1% (< 1×10-3), the patient will be enrolled in the trial and receive consolidation and maintenance treatment according to protocol.

Consolidation - CYCLE 1 Early consolidation chemotherapy that the patients will receive in the first cycle (21 days) consists of: dexamethasone 20 mg/m2 per day, PO or IV days 1-5, 10 mg/m2 per day, PO or IV day 6, 5 mg/m2 per day, PO or IV day 7, 2.5 mg/m2 per day, PO or IV day 8, Vincristine 1.5 mg/m2 per day, IV (maximum 2 mg) days 1 and 8, Methotrexare 3g/m2, IV in 24 hours, E. coli L-asparaginase (L-ASP) (Kidrolase®): 20,000 IU/m2, IV, day 3,Triple intrathecal therapy day 1.

Consolidation - CYCLE 2

Early consolidation chemotherapy that the patient will receive in the second cycle (21 days) consists of:

* Dexamethasone:

  * 20 mg/m2 per day, PO or IV days 1-5.
  * 10 mg/m2 per day, PO or IV day 6.
  * 5 mg/m2 per day, PO or IV day 7.
  * 2.5 mg/m2 per day, PO or IV day 8.
* ARA-C:

  - 2 g/m2 every 12 hours, over 3 hours, days 1 and 2. Halve the ARA-C for patients over 50 years of age.
* E. coli L-asparaginase (L-ASP) (Kidrolase®): 20,000 IU/m2, IV, day 3. Halve the dose for patients over 50 years of age as the toxicity of any type of ASP increases with age.
* Triple intrathecal therapy day 4 (administered that day to keep the intrathecal therapy separate from the high-dose ARA-C).

Consolidation - CYCLE 3 In the third early consolidation cycle, the investigational drug blinatumomab will be administered.

* Blinatumomab 28 μg/day as a continuous infusion, IV over 4 weeks.
* Triple intrathecal therapy day 1.

Late consolidation Two weeks after completing the blinatumomab treatment, in the case of MRD < 0.01% (< 1×10-4), patients will receive 2 blocks of intensive chemotherapy (identical to those in early consolidation), separated by 3 weeks, followed by a treatment cycle with blinatumomab, the investigational medicinal product, for 4 weeks.

After administering late consolidation therapy, a bone marrow study will be conducted. In the case of MRD < 0.01% (< 1×10-4), the patient will receive maintenance treatment. If this MRD level is not achieved, the patient will be withdrawn from the study and undergo a haematopoietic stem cell transplantation, according to routine clinical practice at Spanish sites.

The maintenance therapy that patients will receive in this phase of the trial will consist of continuous chemotherapy administration (mercaptopurine and methotrexate) with reinductions for up to one year from CR

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 18 to 55 years of age, both inclusive.
* Patients with Philadelphia chromosome-negative or BCR-ABL-negative, CD19-positive ALL, with high-risk characteristics. The definition of high-risk ALL implies the presence of one or more of the following factors: Aged 30-55 years; Leukocytes > 30×109/l in B-precursor ALL; Any of the following cytogenetic or molecular abnormalities: 11q23 abnormalities, or proven MLL rearrangement; Complex karyotype (more than 5 chromosome abnormalities); Pro-B ALL, regardless of the number of leukocytes.
* Previous treatment according to routine clinical practice in Spanish centres, in accordance with the PETHEMA protocol for patients with high-risk ALL (ALL-AR-11), in complete remission (MRD < 0.1%) (< 1×10-3) centralised assessment through flow cytometry) after induction therapy.
* ECOG < 2.
* Ability to understand the study and willingness to sign the written informed consent form

Exclusion Criteria:

* Philadelphia chromosome-positive (Ph+) ALL.
* Burkitt's leukaemia (mature B phenotype) according to the WHO classification.
* T-cell ALL.
* B-precursor ALL with high-risk characteristics and MRD ≥ 0.1% (≥ 1×10-3) after receiving induction chemotherapy.
* Previous history or presence of a clinically significant disease of the central nervous system (CNS): epilepsy, seizures, paresis, aphasia, stroke, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, psychosis.
* Presence or history of an autoimmune disease potentially affecting the CNS.
* Radiotherapy in the 2 weeks prior to starting treatment with blinatumomab.
* Immunotherapy (e.g., rituximab) within 4 weeks prior to starting treatment with blinatumomab.
* Any investigational product for leukaemia in the 4 weeks prior to starting treatment with blinatumomab.
* Treatment with any investigational medicinal product after signing the informed consent form.
* Candidate patient for allogeneic haematopoietic stem cell transplantation (HSCT) at the time of enrolment.
* Known hypersensitivity to human immunoglobulins or to any component of the investigational product.
* Abnormal laboratory values: AST (SGOT) and/or ALT (SGPT) and/or alkaline phosphatase ≥ 5 ULN;total bilirubin ≥ 1.5 ULN (unless related to Gilbert's syndrome or Meulengracht's disease); Creatinine ≥ 1.5 ULN; Estimated creatinine clearance < 50 ml/min; Haemoglobin ≥ 9 g/dl (transfusion permitted).
* History of malignant disease other than ALL in the 5 years prior to starting treatment with blinatumomab, with the exception of basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix.
* Active uncontrolled infection, or any other concurrent disease or medical condition considered to interfere with the conduct of the study as per the investigator's discretion.
* HIV infection or chronic hepatitis B virus (HBsAg positive) or hepatitis C virus infection (anti-HCV positive).
* Pregnant or breast-feeding women.
* Women of childbearing potential who are not willing use an effective method of contraception during their participation in the study and for at least 3 months thereafter. Men who are not willing to take measures to prevent their partner from becoming pregnant during their participation in the study and for at least 3 months thereafter.
* Prior treatment with blinatumomab.
* Patients who do not want or are unable to meet the protocol requirements

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2018-06-30 (Actual); Primary Completion 2019-12-24 (Actual); Study Completion 2022-03-09 (Actual)

PRIMARY OUTCOMES:
To assess the reduction rate of the Minimal residual disease determined by Multiparametric flow cytometry | 1 year
  To assess the reduction rate of the MRD determined by MFC, after early consolidation following the inclusion of blinatumomab administered during the early consolidation phase in patients ≤ 55 years of age with high-risk Philadelphia chromosome-negative (Ph-) acute lymphoblastic leukaemia (ALL) with MRD < 0.1% (< 1×10-3) after induction therapy.

CONTACTS AND LOCATIONS:
Locations (12):
- Spain (12):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital ICO Hospitalet, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - . Hospital Clínico Universitario Virgen de la Victoria, Málaga
  - Hospital Central de Asturias, Oviedo
  - Hospital Clinico Universitario de Salamanca, Salamanca
  - C.H.U, de Santiago, Santiago de Compostela
  - H. Virgen Del Rocio, Seville
  - Hospital Universitario y Politécnico la Fe, Valencia

IPD SHARING:
Plan to Share IPD: Undecided